CLINICAL TRIAL: NCT05630131
Title: Pilot Study to Evaluate the Role for Circulating Tumor DNA (ctDNA) in Monitoring Subjects With Muscle-invasive Bladder Cancer Treated With Trimodality Therapy
Brief Title: ctDNA in Subjects With Muscle-invasive Bladder Cancer Treated With Trimodality Therapy
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC2208
Record Dates: First submitted 2022-11-17; First posted 2022-11-29 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Bladder Cancer; Muscle-Invasive Bladder Carcinoma
Keywords: circulating tumor DNA; biospecimen; surgery; radiotherapy; chemotherapy; trimodality
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — urine and blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this prospective biospecimen collection study is to evaluate the feasibility of measuring circulating tumor DNA (ctDNA) in subjects with muscle-invasive bladder cancer (MIBC) treated with trimodality therapy consisting of a maximal transurethral resection of bladder tumor followed by radiation and concomitant chemotherapy.

Cancer cells have unique genes that determine the characteristics of tumors, such as how they will respond to different treatments. The tumor tissue will be used to determine the genes present in cancer cells. Tumor cells sometimes release fragments of DNA into the blood or urine (circulating tumor DNA or ctDNA) and measuring levels of ctDNA may be a way to monitor cancer and predict to determine which treatment works better and what will be the outcome of cancer.

Urine, blood, and tumor tissue are called biospecimens. Biospecimens can help researchers understand how the human body works. Researchers may develop new tests to monitor diseases or new ways to treat diseases. Plasma and urine specimens will be collected before, during, and after the standard-of-care treatment.

This study will estimate the feasibility of collecting plasma ctDNA detection in subjects with MIBC. If this information can be successfully collected and processed, the usefulness of ctDNA to predict tumor response to certain kinds of treatment or disease progression will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent was obtained to participate in the study and HIPAA authorization for the release of personal health information.
2. A diagnosis of Muscle-invasive Bladder Cancer with a plan to treat it with surgery, radiation, and chemotherapy
3. Subjects are willing and able to comply with study procedures based on the judgment of the investigator.

Exclusion Criteria:

All subjects must not meet any of the following exclusion criteria prior to enrollment to participate in this study:

1. Any serious medical or psychiatric disorder that would interfere with the subject's ability to give informed consent.
2. Incarcerated individuals.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: University of North Carolina Patients
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2025-08-02 (Actual); Study Completion 2025-08-02 (Actual)

PRIMARY OUTCOMES:
Feasibility of cell-free plasma ctDNA collection | Up to 2 years
  The feasibility of cell-free plasma ctDNA collection will be estimated by the percentage of specimens that yield a ctDNA result.

SECONDARY OUTCOMES:
Feasibility of urine ctDNA collection | Up to 2 years
  The feasibility of urine ctDNA collection will be estimated by the percentage of specimens that hat yield a ctDNA result.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew I Milowsky, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- North Carolina Cancer Hospital (UNC), Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with other researchers.

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials